CLINICAL TRIAL: NCT02265913
Title: Comparative Safety and Efficacy of Two Antiviral Treatments in the Treatment of Recurrent Herpes Simplex Labialis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-NY-14-008
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Herpes Labialis
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Product (Experimental): acyclovir cream
  Interventions: Drug: Acyclovir 5 percent (Perrigo)
- Reference Product (Active Comparator): acyclovir cream
  Interventions: Drug: Acyclovir 5 percent (Reference)
- Placebo Product (Placebo Comparator): Placebo cream
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: Acyclovir 5 percent (Perrigo)
  Other Names: Perrigo product
  Arms: Test Product
Drug: Acyclovir 5 percent (Reference)
  Other Names: Reference Listed Drug Product
  Arms: Reference Product
Drug: Placebo cream
  Arms: Placebo Product

SUMMARY:
To compare safety and efficacy of Perrigo's antiviral drug product compared to an FDA approved antiviral drug product in the treatment of cold sores.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent/assent
2. Immunocompetent male or non-pregnant females, >12 years old, with limited, non-life-threatening, recurrent herpes simplex labialis.
3. Subjects must have at least 3 recurrences of herpes simplex labialis per year for the past two years.
4. Females of childbearing potential willing to use an acceptable form of birth control.
5. Subjects must be in general good health with no clinically significant disease that might interfere with the study evaluations in the opinion of the investigator.
6. Subjects must be willing and able to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Females who are pregnant or nursing, are not using or does not agree to use an acceptable form of contraception during the study, or who intends to become pregnant during the study.
2. The use of antiviral therapies in various forms for a given period of time prior to screening and study medication application.
3. Candidate for or previous use of parenteral antiviral treatment or prophylactic antiviral therapy for their recurrent herpes simplex labialis.
4. Recently received an organ transplant.
5. Subjects who are immunocompromised, HIV positive or who have any immune-system disorders.
6. Recent major change in immune system status that could seriously affect the clinical manifestations of herpes simplex labialis and need for treatment in the opinion of the investigator.
7. Subjects with known or suspected history of a clinically significant systemic disease, unstable medical disorders, life-threatening disease or current malignancies.
8. Subjects with a current episode of herpes simplex labialis that has not completely healed.
9. Presence of any facial skin condition or excessive facial hair that may interfere with diagnosis, assessment, and/or healing ability.
10. History of herpes keratitis.
11. Subject has a history of hypersensitivity or allergy to any ingredient in the drug product.
12. History of unresponsiveness to topical acyclovir therapy.
13. Participation in any other clinical study or who have received treatment with any investigational drug or device within 30 days prior to screening.
14. Subjects who have previously enrolled in this study.
15. Subjects who have received any local medication in the target area during the 2 weeks prior to both enrollment/screening and Day 1 (Visit 2).
16. Subjects who have been treated with immunosuppressive medication therapy within 8 weeks prior to the study both enrollment/screening and Day 1 (Visit 2).
17. Subject consumes excessive alcohol, abuses drugs, or has a condition that could compromise the subject's ability to comply with study requirements in the investigator's opinion.
18. Use of tanning booths, sun lamps, or excessive exposure to the sun for up to 21 days from initiating study medication
19. Subjects using immunostimulators, dye-light therapy, or psoralen therapy within 30 days prior to study medication initiation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4076 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quality Clinical Research Inc, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product: acyclovir cream
  Acyclovir 5 percent (Perrigo)
- Reference Product: acyclovir cream
  Acyclovir 5 percent (Reference)
Period: Overall Study
Arm/Group | Test Product | Reference Product | Placebo Product
Started | 1357 | 1361 | 1358
Completed | 793 | 810 | 813
Not Completed | 564 | 551 | 545

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Placebo Product | Total
Number analyzed (Participants) | 1357 | 1361 | 1358 | 4076
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (15.05) | 43.9 (15.20) | 43.3 (14.99) | 43.7 (15.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 900 | 915 | 902 | 2717
  Male | 457 | 446 | 456 | 1359
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 278 | 297 | 300 | 875
  Not Hispanic or Latino | 1079 | 1064 | 1057 | 3200
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 4 | 16
  Asian | 9 | 12 | 9 | 30
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 3 | 9
  Black or African American | 294 | 284 | 244 | 822
  White | 1025 | 1037 | 1078 | 3140
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 20 | 19 | 20 | 59

OUTCOME MEASURES:

1. Primary Outcome: Lesion Healing
Description: Time to complete healing of lesions measured in hours from the time of first dosing
Time Frame: up to 21 days
Population: per protocol population
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Test Product: acyclovir cream: Acyclovir 5 percent (Perrigo)
- Reference Product: acyclovir cream: Acyclovir 5 percent (Zovirax)
- Placebo Product: vehicle of the test product cream
Arm/Group | Test Product | Reference Product | Placebo Product
Number analyzed (Participants) | 633 | 652 | 641
hours | 107.47 (80.660) | 110.08 (82.840) | 112.41 (83.467)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Equivalence — provides 85% of success; Fieller's method; Equivalence ratio = 98.0, 90% CI 2-sided [92 to 105]

ADVERSE EVENTS:
Time Frame: Up to 21 days
Arm/Group | Test Product | Reference Product | Placebo Product
All-Cause Mortality (participants affected / at risk) | 0/1357 | 0/1361 | 0/1358
Serious Adverse Events (participants affected / at risk) | 2/1357 | 4/1361 | 0/1358
Other Adverse Events (participants affected / at risk) | 0/1357 | 0/1361 | 0/1358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=1357) | Reference Product (N=1361) | Placebo Product (N=1358)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Worsening Of Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Kidney Stone (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Right Forearm Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT02265913/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT02265913/SAP_001.pdf